CLINICAL TRIAL: NCT02817282
Title: Compliance With Hand Hygiene in Nursing Homes: Go for a Sustainable Effect (CHANGE)
Acronym: CHANGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: National Institute for Public Health and the Environment (RIVM) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 50-53000-98-113
Record Dates: First submitted 2016-02-22; First posted 2016-06-29 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-07

CONDITIONS: Infectious and Communicable Diseases
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hand hygiene implementation strategy (Other): The implementation strategy will be tested in a stepped wedge cluster randomized trial which is based on a random sequential roll-out of the CHANGE implementation strategy to all participating NHs (n=20) for comparison. All groups (hence all NHs) start with the control situation (no CHANGE implementation activities) at the beginning of the study. At each time point, a new group of five NHs crosses over from the control situation to the implementation situation. Each group will start the implementation phase of 4 months at a different time point, directly after one of the measurements periods (Point of Time (PT) 0, PT1, PT2, PT3, PT4, PT5). The time point a group crosses over is randomized (over the groups).
  Interventions: Other: Hand hygiene implementation strategy

INTERVENTIONS:
Other: Hand hygiene implementation strategy — Implementation strategy: Individual oriented activities. Education based on the different determinants influencing HCWs' behavior. Reminders for supporting the actual performance of HH; by distributing posters. Performance feedback for awareness. Goal setting will be encouraged and the feedback will be used to help HCWs evaluate their success and determine how they could best adapt their behavior in order to reach their goal. Organisational oriented activities. Products and facilities: The physical environment will be adapted by improving the availability of hand based hand rub. Team-oriented activities; The social environment will be adapted by training at a group and individual level, to improve social and descriptive norms. Positive role models will be stimulated through this training.

SUMMARY:
Hand hygiene (HH) appears to be a simple, non-complex procedure to prevent healthcare-associated infections (HAIs), implementation in daily routine is difficult. The residential setting and specific population pose challenges to optimal HH compliance. This study aims to develop and to evaluate an evidence based multi-component implementation strategy aimed at the promotion of HH in Dutch nursing homes(NHs). A strategy to improve HH compliance in Dutch NHs will be developed. This strategy addresses the specific barriers and facilitators of NHs' infrastructure, healthcare workers (HCWs) and socio-cultural setting. The strategy will be tested in a stepped wedge cluster randomized design which is based on a random sequential roll-out of the implementation strategy to all participating NHs (n=20) for comparison. Data are collected during six consecutive four month periods with an initial baseline period for all NHs.

During each period 1200 opportunities for HH are observed, using the gold standard of direct and unobtrusive observations, according to the Five Moments for HH of the World Health Organization. HAIs incidence densities, collected in the sentinel surveillance network for infectious diseases in nursing homes (SNIV), will be evaluated in parallel.

A multi component implementation strategy, combining activities aimed at individual HCWs, teams and the organization will be used. The individual level includes education, skills, action planning, reminders and feedback. The team level includes activities that focus on social influence, strengthening of leadership by gaining active commitment and initiative of ward management. The organizational level addresses the structural context and institutional management support.

To assess the cost implications of the CHANGE strategy, an economic evaluation will be conducted from a healthcare perspective. The cost-effectiveness of improved HH, defined here as the costs for the CHANGE strategy minus less costs for treating infections, divided by the difference between HAIs before and after the intervention period, will be calculated. A process evaluation will be performed during and after the intervention to investigate the feasibility of the implementation strategy and to illuminate the mechanisms and processes responsible for the results and their variation within the NHs.

DETAILED DESCRIPTION:
Sub study I: In an observational study, current HH compliance will be assessed in the participating NHs, by using direct but unobtrusive observation. The primary outcome is the percentage of opportunities at which HH is performed in accordance with the WHO guideline.

Direct observation will be used as this is considered the gold standard and the most reliable method for assessing compliance rates. Direct observation makes it possible to examine and quantify the required moments for HH and assess the quality of practice.

Strigley et al. showed that HH compliance rates were approximately threefold higher within eyesight of an auditor compared with when no auditor was visible. Therefore, observations will be performed unobtrusively to diminish the Hawthorne effect-the possibility that HCWs modify their HH behavior in response to the fact that they know they are being studied. At the beginning of each observation period, HCWs will be informed that the observers conduct research on patient safety errors, but not that HH is monitored. Only the director of the ward will be informed about the real purpose of the observations. This method of observation was feasible in previous projects and is currently the World Health Organisation (WHO)-recommended standard for evaluating HH.

Sub study II: Barriers and facilitators in performing HH. To develop a successful HH strategy in NHs, information is needed on the behavioral determinants of HH compliance. In line with a study by Grol among doctors and nurses in hospitals and nursing homes, identified barriers are related to the individual HCW (e.g. not convinced of the evidence, working routines); the social context within the team (e.g. no mutual accountability and control, no leadership); and the healthcare organisation (high workload, insufficient facilities). Perceived barriers to adherence with HH guidelines also include skin irritation caused by HH agents, interference with HCWs' relationships with patients, patient needs perceived as a priority over HH, and the lack of scientific information showing that HH prevents cross-infection. Erasmus et al. found also that negative role models, poor accessibility of materials and a poor social culture hamper good HH. Finally, a recent Cochrane review of the effectiveness of 'tailored' strategies gave a foundation to the assumption that strategies for change are more effective if they deliberately address identified barriers.

In this study the barriers and facilitators are experienced in performing HH in Dutch NHs will be explored. From the literature on barriers to guideline implementation combined with a literature study on barriers in performing HH, a barriers questionnaire was previously developed and used in the Helping Hands study. To ensure that the questionnaire contains all possible barriers that can be experienced in the NH setting, focus group discussions with HCWs in NHs will be performed. Newly mentioned barriers will be included in the questionnaire. Next, a questionnaire study will be performed among a random sample of all professionals, with a minimum of 25 in the participating NH to identify the most frequently experienced barriers among professionals.

Sub study III: development of HH implementation strategy individual oriented activities. Education will be based on the different determinants influencing HCWs' behavior. Reminders for supporting the actual performance of HH will be used by distributing posters that emphasize the importance of HH, particularly alcohol-based hand disinfection.

Performance feedback is an effective tool to increase awareness, and has often been effective in improving HH for short periods. Different mediums will be used for communicating the feedback of HH performance of the own unit in comparison to other experimental units. The results will also be discussed in staff meetings. This element will be embeded into pre-existing work routines. Goal setting will be encouraged and the performance feedback will be used to help HCWs evaluate their success and determine how they could best adapt their behavior in order to reach their goal.

Planning for improvement; during HCWs' busy day to day activities will be increased by making action plans (implementation intentions), as part of the education program in which HCWs will be assisted in making concrete plans and solutions to the everyday problems they encounter concerning HH, using if-then plans (web based and/or in groups). Concretely it will involve formulating plans how and when they intend to perform hand hygiene (i.e. when washing a resident, first walk to the hand alcohol dispenser). This type of intervention has shown promising results in creating new habits and changing fixed behaviours in other areas of public health.

Organisational oriented activities Products and facilities: The physical environment will be adapted by screening and improving the availability of hand based hand rub.

Team-oriented activities:The social environment will be adapted by training at a group and individual level, to improve social and descriptive norms. Positive role models will be stimulated through this training, and particularly senior HCWs will be encouraged to improve their behavior as role models. The intervention will be delivered in two interactive team sessions during a period of 6 months. The first 1,5-h team session start with presenting and discussing current the team performance on HH. Team members explore their HH behavior, analyse barriers and facilitators and formulate improvement activities. Next, team members develop a clear set of behavior and communication expectations to address each other in case of inappropriate HH. The meeting ends with commitment of all team members to achieve a substantial increase in HH compliance. During the second session, the ward manager will present the HH compliance rates of the previous period. Team members discuss questions like: Is the goal achieve? What improvements have been implemented? How to maintain the improved behavior? What went wrong and what to do about it? Next, attention will be focused at maintenance of the achieved results.

Implementation of CHANGE: In order to increase the success of implementation, an extensive strategy will be put in place prior to the start of the intervention period. In each NH contact persons will be appointed: the coordinating Infection Control Practitioner (ICP). With them the roll-out of the CHANGE package in their NH will be discussed. At the start of the intervention a kick-off meeting will be planned in the participating NH. HCWs will be instructed as to how they can signal when a component of the intervention is interfering with their work activities, so that effective measures to solve these problems can be set in motion swiftly. Education and team training will be timely planned and integrated in regular work meetings and in existing educational courses. The implementation phase per NH will last 4 months. During a period of two years, all NHs will receive the implementation strategy.

Sub study IV evaluation of HH implementation strategy. The implementation strategy will be tested in a stepped wedge cluster randomized trial which is based on a random sequential roll-out of the CHANGE implementation strategy to all participating NHs (n=20) for comparison. All groups (hence all NHs) start with the control situation (no CHANGE implementation activities) at the beginning of the study. At each time point, a new group of five NHs crosses over from the control situation to the implementation situation. Each group will start the implementation phase of 4 months at a different time point, directly after one of the measurements periods (Point of time (PT)0, PT1, PT2, PT3, PT4, PT5). The time point a group crosses over is randomized (over the groups). Randomization will be computer generated by an independent statistician when recruitment of clusters is complete. By the end of the two year study period, all groups (hence all NHs) will have received the CHANGE implementation strategy.

Sub study V: Exploratory economic evaluation. Costs of HAIs are high and HH is an effective measure in reducing infections. It is estimated that 15 to 30% of all HAIs can be prevented by avoiding cross-transmission of micro-organisms on the hands of HCWs. An improvement in HH compliance has potential to lead to substantial health care cost savings. Therefore, strategies that focus on increasing adherence to effective HH guidelines are likely to be cost-effective. To date, little is known about the costs induced by non-compliance to HH in NHs. To assess the cost implications of inadequate HH, an economic evaluation will be conducted from a healthcare perspective. The economic evaluation will be performed in accordance with the Dutch guidelines, the general principles of cost-effectiveness analysis in healthcare. In the CHANGE implementation strategy the HH compliance in the participating NHs will increase and subsequently will lead to a decrease in the incidence of HAIs. Data will be collected on healthcare use for HAIs that are monitored in the participating NHs.

For the calculation of potential cost savings due to less infections, the use of antibiotics and other drugs, contact isolation precautions, extra consultations of the elderly care physician, diagnostic tests, extra medical care, hospital transportation and hospital admission will be registered . Weekly, participating NHs register the incidence of HAIs. This registration makes it possible to compare the incidence of infections before the intervention period with the incidence of infections during and after the intervention period. This allows for the possibility to calculate the cost-effectiveness of improved HH, defined here as the costs for the CHANGE strategy minus less costs for treating infections, divided by the difference between HAIs before and after the intervention period.

Sub study VI: process evaluation. A process evaluation will be performed during and after the intervention to investigate the feasibility of the implementation strategy and to illuminate the mechanisms and processes responsible for the results and their variation within the NHs. For this purpose, the different implementation activities and the participation level of the HCWs in order to determine the correlation between the implementation effect (i.e., results of our implementation strategy on HH compliance) and adherence to the implementation strategy (i.e., degree of implementation) will be registered. To understand the success -or lack of success- of the implementation strategy, the evaluation will use three sets of measures that will be related to the effects on HCWs' HH compliance: adherence to the improvement strategy, contextual factors, and HCWs' experiences with strategy components. Information on adherence to the improvement strategy and on contextual factors will be collected using a wide range of methods, including: observations, a NH structure survey, structured logbooks of coaches and researchers' field notes of group meetings etc. For example, participation in the implementation activities will be monitored closely, by documenting participation regarding all activities: e.g. who participated in an educational meeting, who read his/her individual feedback report etc. This information is not only crucial for understanding the result of implementation strategy, but also for providing basic data for the economic evaluation of the improvement activities. Information on HCWs' experiences with strategy components will be collected by such information is not only crucial for understanding the result of implementation strategy, but will also be measured to, if necessary, adapt the strategy to make it more acceptable and effective for future users of the strategy.

ELIGIBILITY:
Inclusion Criteria:

Nursing homes has to join the incidence registration of the national network SNIV (Surveillance Network of Infectious diseases in Nursing homes)

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Hand hygiene compliance | two year
  Data are collected during six consecutive periods of 4 month each (Point of time (PT) 0,PT1,PT2,PT3,PT4 and PT5); 1200 opportunities for HH compliance in the NH's are observed during each time period. At each data collection period (PT0-PT5) 60 opportunities for HH compliance, in 12-15 HCWs, per NH will be observed

SECONDARY OUTCOMES:
Healthcare associated infections | 2 years
  The incidence of HAIs in the participating NHs will be collected through the routine SNIV surveillance. In this surveillance network, infections are reported weekly through a web-based application. Only new episodes of an infection are registered

CONTACTS AND LOCATIONS:
Overall Officials: Marlies Hulsher, Prof Dr, Principal Investigator — UMC Radboud

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Teerenstra S, Taljaard M, Haenen A, Huis A, Atsma F, Rodwell L, Hulscher M. Sample size calculation for stepped-wedge cluster-randomized trials with more than two levels of clustering. Clin Trials. 2019 Jun;16(3):225-236. doi: 10.1177/1740774519829053. Epub 2019 Apr 24. PMID 31018678